CLINICAL TRIAL: NCT06564038
Title: A Phase I/II Open-Label Multi-Centre Master Protocol to Evaluate the Safety and Efficacy of AZD0486 Monotherapy or in Combination With Other Anticancer Agents in Participants With Mature B-Cell Malignancies
Brief Title: A Study of AZD0486 Monotherapy or in Combination With Other Anti-Cancer Agents for Mature B-Cell Malignancies
Acronym: Soundtrack-E
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7407C00001; 2024-515034-33-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukaemia; Small Lymphocytic Lymphoma; Mantle-cell Lymphoma; Large B-cell Lymphoma; B-cell Non-Hodgkin Lymphoma
Keywords: IgG4 fully human CD19xCD3 bispecific T-cell engager; B cell lymphoma; Subcutaneous; AZD0486; Acalabrutinib; Prednisone; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Surovatamig
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, B-Cell | interventions — Prednisone; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Substudy 1 (RR CLL/SLL): Cohort 1A (AZD0486 Monotherapy) (Experimental): Participants will receive AZD0486 monotherapy as subcutaneous (SC) injection.
  Interventions: Drug: AZD0486
- Substudy 1 (RR CLL/SLL): Cohort 1B (AZD0486 + Acalabrutinib) (Experimental): Participants will receive AZD0486 as SC injection. Participants will receive acalabrutinib tablet orally twice daily.
  Interventions: Drug: AZD0486; Drug: Acalabrutinib
- Substudy 1 (RR CLL/SLL): Cohort 1C (AZD0486 Monotherapy) (Experimental): Participants will receive AZD0486 monotherapy as intravenous (IV) infusion.
  Interventions: Drug: AZD0486
- Substudy 2 (RR MCL): Cohort 2A (AZD0486 Monotherapy) (Experimental): Participants will receive AZD0486 monotherapy as SC injection.
  Interventions: Drug: AZD0486
- Substudy 2 (RR MCL): Cohort 2C (AZD0486 Monotherapy) (Experimental): Participants will receive AZD0486 monotherapy as IV infusion.
  Interventions: Drug: AZD0486
- Substudy 3 (LBCL): AZD0486 + R-CHOP (Experimental): Participants will receive AZD0486 as IV infusion in combination with R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) chemotherapy.
  Interventions: Drug: AZD0486; Drug: Prednisone (or equivalent); Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin

INTERVENTIONS:
Drug: AZD0486 — AZD0486 will be administered as either SC injection or IV infusion.
  Other Names: TNB-486; Surovatamig
Drug: Prednisone (or equivalent) — Prednisone (or equivalent) will be administered either oral or IV infusion as per standard of care.
  Arms: Substudy 3 (LBCL): AZD0486 + R-CHOP
Drug: Rituximab — Rituximab will be administered as IV infusion as per standard of care.
  Arms: Substudy 3 (LBCL): AZD0486 + R-CHOP
Drug: Cyclophosphamide — Cyclophosphamide will be administered as IV infusion as per standard of care.
  Arms: Substudy 3 (LBCL): AZD0486 + R-CHOP
Drug: Vincristine — Vincristine will be administered as IV infusion as per standard of care.
  Arms: Substudy 3 (LBCL): AZD0486 + R-CHOP
Drug: Doxorubicin — Doxorubicin will be administered as IV infusion as per standard of care.
  Arms: Substudy 3 (LBCL): AZD0486 + R-CHOP
Drug: Acalabrutinib — Acalabrutinib will be administered orally
  Arms: Substudy 1 (RR CLL/SLL): Cohort 1B (AZD0486 + Acalabrutinib)

SUMMARY:
The purpose of this study is to assess the safety and efficacy of AZD0486 administered as monotherapy or in combination with other anticancer agents in participants with hematological malignancies.

DETAILED DESCRIPTION:
This is open-label, multi-center study to evaluate the safety and preliminary efficacy of AZD0486 administered as monotherapy and in combination with other anticancer agents in participants with mature B-cell hematologic malignancies.

This master study currently includes 3 substudies and each substudy focusing on a defined population:

Substudy 1: Relapsed/refractory (R/R) Chronic lymphocytic leukaemia (CLL)/ Small lymphocytic lymphoma (SLL) Substudy 2: R/R Mantle-cell lymphoma (MCL) Substudy 3: Large B-cell lymphoma (LBCL) or R/R B-cell non-Hodgkin lymphoma (B-NHL) (not applicable to US)

The study will have the following sequential periods:

1. Screening period of 28 days
2. Treatment period
3. Follow-up period

ELIGIBILITY:
Inclusion Criteria:

Master Inclusion Criteria applicable to all substudies:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Contraception use during treatment and at least 90 days after final dose.
* Confirmed CD19 expression if prior anti-CD19 therapy.

Substudy 1 Specific Inclusion Criteria:

* Participants with CLL must require treatment according to the international workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria.
* SLL: at least 1 measurable site per Lugano.
* Absolute lymphocytes <10,000.
* Cohort 1A and 1C: at least 2 prior lines of systemic therapy for CLL/SLL.
* Cohort 1B: at least 1 prior line of therapy and is bruton tyrosine kinase inhibitor (BTKi)-sensitive.

Substudy 2 Specific Inclusion Criteria:

* MCL diagnosis per WHO.
* Clinical Stage II, III, or IV by Ann Arbor Classification.
* At least 1 measurable site per Lugano.
* ALC < 10,000.
* Cohort 2A and 2C: Relapse or progressed after 2 or more lines of therapy including BTKi.

Substudy 3 Specific Inclusion Criteria:

* Large B-cell lymphoma per WHO 2022.
* R/R B-NHL after at least 1 prior line of therapy.
* International Prognostic Index (IPI) 2-5.
* At least 1 measurable site as per Lugano.
* Left ventricular ejection fraction (LVEF) >50%.
* Contraception at least 90 days after last dose of AZD0486 or 4 months after last dose of vincristine, and 6 months after the last dose of cyclophosphamide, or doxorubicin.

Exclusion Criteria:

Master Exclusion Criteria applicable to all substudies:

* Central nervous system (CNS) lymphoma.
* Surgery within 14 days of study drug.
* Clinically significant cardiovascular (CV) disease.
* Unresolved Grade >2 AEs from prior anticancer therapy (except alopecia or fatigue).
* Any anticancer therapy within 5 half-lives or 21 days (whichever is shorter) prior to treatment.
* Radiation therapy within 28 days.
* Prior CAR T-cell therapy or autologous-haematopoietic stem cell transplant (HSCT) within 12 weeks or prior T-cell engager (TCE) within 8 weeks.
* Prior Grade > 3 cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity syndrome (ICANS) event.
* Prior allogeneic HSCT or solid organ transplantation within 24 weeks of starting Cycle 1 Day 1.

Substudy 1 Specific Exclusion Criteria:

* CLL transformation to more aggressive lymphoma.
* Cohort 1B: bleeding diathesis, CYP3A inhibitor or inducer, history of ICH or stroke within 24 weeks, GI malabsorption, receiving vitamin K antagonist.

Substudy 3 Specific Exclusion Criteria:

* Mediastinal grey-zone lymphoma, Burkitt, Richter's transformation, primary effusion large B-cell lymphoma (LBCL).
* Cumulative dose of anthracycline >150 mg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events, Serious Adverse Events and Adverse Events of Special Interest | Up to 6 years 4 months
  Safety and tolerability of AZD0486 as monotherapy and in combination with other anticancer agents across mature B-cell malignancies.
Number of Participants with Dose Limiting Toxicity (DLTs) | Up to 2 months
  Safety and tolerability of AZD0486 as monotherapy and in combination with other anticancer agents across mature B-cell malignancies.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 6 years 4 months
  ORR is defined as percentage of participants achieving either a partial response (PR) or complete response (CR) based on response criteria for International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 and Lugano 2014 assessed by investigator (substudy 1) and percentage of participants achieving CR as best response based on Lugano 2014 Response Criteria by investigator assessment (substudies 2 and 3).
Complete Response (CR) Rate | Up to 6 years 4 months
  CR rate is defined as percentage of participants achieving CR as best response based on response criteria for iwCLL 2018 and Lugano 2014 assessed by investigator (substudy 1) and percentage of participants achieving CR as best response based on Lugano 2014 Response Criteria by investigator assessment (substudies 2 and 3).
Duration of Response (DoR) | Up to 6 years 4 months
  DoR is defined as time from the date of first documented response until date of documented progression based on response criteria for iwCLL 2018 and Lugano 2014 assessed by investigator, relapse or death (substudy 1) and time from the date of first documented response until date of documented progression based on Lugano 2014 Response Criteria by investigator assessment, relapse or death (substudies 2 and 3).
Maximum Observed Concentration (Cmax) | Up to 90 days after last dose
  The PK (Cmax) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Area Under the Concentration-time Curve (AUC) | Up to 90 days after last dose
  The PK (AUC) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Minimum Observed Concentration (Cmin) | Up to 90 days after last dose
  The PK (Cmin) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Time to Reach Maximum Concentration (Tmax) | Up to 90 days after last dose
  The PK (Tmax) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Trough Plasma Concentration (Ctrough) | Up to 90 days after last dose
  The PK (Ctrough) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Half Life (t1/2) of AZD0486 | Up to 90 days after last dose
  The PK (t1/2) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Clearance (CL) of AZD0486 | Up to 90 days after last dose
  The PK (CL) of AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.
Number of Participants with Anti-drug Antibody (ADA) for AZD0486 | Up to 90 days after last dose
  The incidence of immunogenicity of SC AZD0486 as monotherapy and in combination with other anti-cancer agents will be evaluated.

CONTACTS AND LOCATIONS:
Locations (56):
- United States (11):
  - Research Site, Boston, Massachusetts
  - Research Site, Hackensack, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Heidelberg
  - Research Site, Melbourne
  - Research Site, Nedlands
- China (5):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Jinan
  - Research Site, Tianjin
  - Research Site, Zhengzhou
- Czechia (3):
  - Research Site, Ostrava - Poruba
  - Research Site, Prague
  - Research Site, Praha 2 - Nové Město
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Copenhagen
  - Research Site, Odense C
- France (5):
  - Research Site, Clermont-Ferrand
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Saint-Cloud
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Cologne
  - Research Site, Kiel
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Würzburg
- Italy (2):
  - Research Site, Bologna
  - Research Site, Milan
- Japan (3):
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Nagoya
- South Korea (2):
  - Research Site, Busan
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Palma de Mallorca
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (4):
  - Research Site, Derriford
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via there quest portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/